CLINICAL TRIAL: NCT06730230
Title: Partners in Control, Phase II: Using Remote Monitoring Technology With Community Health Workers to Support Hypertension Management for Latinx Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-00746; 1R01MD018520-01A1 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Remote Patient Monitoring; Palliative Care

STUDY DESIGN:
Intervention Model Description: With the stepped-wedge design, each clinic will function as a control or "usual care" group prior to the implementation of the intervention. During this period, the clinic will prescribe and treat patients enrolled in the RPM hypertension program using usual protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Latinx patients with uncontrolled hypertension (HTN) (Experimental): Patients will be exposed to the RPM-enabled CHW support, this will be carried out through the step-wedge design, meaning that over the course of the study (~18 months), all clinics will carry out standard HTN care and also have exposure to the intervention (though at varying time intervals).
  Interventions: Behavioral: Remote Patient Monitoring (RPM)-enabled Community Health Worker (CHW) Support

INTERVENTIONS:
Behavioral: Remote Patient Monitoring (RPM)-enabled Community Health Worker (CHW) Support — CHWs will implement RPM by being provided with training modules and implementing electronic health record (EHR) support tools for HTN management.

SUMMARY:
This study seeks to evaluate the impact of a remote patient monitoring (RPM)-specific tech-enabled community health worker workforce on the use of RPM for the management of hypertension among Latinx patients. This study is a step-wedge randomized controlled trial that aims to assess the effectiveness and implementation of RPM-enabled community health workers (CHWs) compared to standard of care RPM hypertension management on blood pressure reduction and evaluate the implementation of the RPM-enabled CHWs for hypertension (HTN) management. The study aims to examine adoption, acceptability, fidelity, cost, sustainability, and equity as outcomes of implementation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Latinx
2. Be fluent in English or Spanish
3. Be age 18 years or older
4. Receiving care at one of the 10 safety-net primary care clinics
5. Have uncontrolled HTN documented in the electronic health record (EHR) on at least two visits in the past year (defined as an average BP ≥ 140/90 mmHg)
6. Have been prescribed at least one anti-hypertensive medication and be non-adherent to their medications, defined as adherence <80% in the preceding 12 months, as determined by prescription orders obtained from the clinic EHR.

Exclusion Criteria:

1. Being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks)
2. Participation in other hypertension-related clinical trials
3. Have significant psychiatric comorbidity or reports of substance abuse (as documented in the EHR)
4. Plan to discontinue care at the clinic within the next 15 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Baseline, Month 18
Change in diastolic blood pressure | Baseline, Month 18

SECONDARY OUTCOMES:
Rate of hypertension control | Month 18
  Outcome measure will be assessed using the National Quality Forum-defined thresholds for controlled/uncontrolled hypertension (BP<140/90 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Devin.Mann@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Devin.Mann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.